CLINICAL TRIAL: NCT05850234
Title: A Phase 1b/2 Study of GC012F (AZD0120), a Chimeric Antigen Receptor T-cell (CAR T) Therapy Targeting CD19 and B-cell Maturation Antigen (BCMA) in Subjects With Relapsed/Refractory Multiple Myeloma
Brief Title: A Study of GC012F (AZD0120), a CAR T Therapy Targeting CD19 and BCMA in Subjects With Relapsed/Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8310C00001; GC012F-CD19/BCMA-001 (Other: Gracell Biopharmaceuticals)
Record Dates: First submitted 2023-04-18; First posted 2023-05-09 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Relapsed/ Refractory Multiple Myeloma
Keywords: Multiple Myeloma, BCMA, CAR
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: GC012F (AZD0120) will be administrated in one infusion
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GC012F (AZD0120) (Experimental): GC012F (AZD0120) will be administrated in one infusion
  Interventions: Biological: GC012F (AZD0120)

INTERVENTIONS:
Biological: GC012F (AZD0120) — GC012F (AZD0120) is a BCMA/CD19 dual CAR product under investigation for the treatment of patients with RRMM.

SUMMARY:
This trial is a phase 1b/2, open-label, multicenter study of GC012F (AZD0120), a CD19/BCMA dual CART-cell therapy, in adult subjects with relapsed/refractory Multiple Myeloma.

DETAILED DESCRIPTION:
For Phase Ib It aims to evaluate the safety, tolerability, pharmacokinetic characteristics, pharmacodynamic effect, immunogenicity in subjects with relapsed/ refractory Multiple Myeloma, and determine the recommended Phase 2 dose of GC012F (AZD0120).

For Phase 2, it aims to evaluate the efficacy, to further characterize the safety of GC012F (AZD0120), pharmacodynamic effect, and immunogenicity, changes from baseline for subject-reported health-related quality of life, overall health status in subjects with relapsed/ refractory Multiple Myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥18 years of age at the time of consent
* Written informed consent in accordance with federal, local, and institutional guidelines
* Have an ECOG performance status of 0 or 1
* Documented diagnosis of MM per IMWG diagnostic criteria
* Received at least three prior MM treatment lines of therapy
* Have received as part of their previous therapy a PI and IMiD and an antiCD38 antibody.
* Have documented evidence of progressive disease by the IMWG criteria.
* Subjects must have measurable disease at screening, as defined by any of the following: serum monoclonal paraprotein (M-protein) ≥1.0g/dL (10 g/L); urine M-protein ≥200 mg/24 h; serum FLC assay: involved FLC level is ≥10 mg/dL (100 mg/L) and serum kappa lambda FLC ratio is abnormal.
* Adequate bone marrow and organ function assessment at screening according to the hematological, hepatic, and renal parameters listed in the CSP

Exclusion Criteria :

* Diagnosed or treated for invasive malignancy other than multiple myeloma, except: Malignancy treated with curative intent and with no known active disease present for ≥2 years before enrollment; or
* Adequately treated non-melanoma skin cancer without evidence of disease.
* The following cardiac conditions:
* New York Heart Association (NYHA) stage III or IV congestive heart failure
* Myocardial infarction or coronary artery bypass graft (CABG) ≤6 months prior to enrollment
* History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration
* History of severe non-ischemic cardiomyopathy
* Received either of the following:
* An allogenic stem cell transplant within 6 months before apheresis. Subjects who received an allogeneic transplant must be off all immunosuppressive medications for 6 weeks without signs of graft-versus-host disease (GVHD).
* An autologous stem cell transplant ≤12 weeks before apheresis
* Known active, or prior history of central nervous system (CNS) involvement or exhibits clinical signs of meningeal involvement of multiple myeloma.
* Plasma cell leukemia at the time of screening (>2.0×109 /L plasma cells by standard differential), Waldenström's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes), or primary AL amyloidosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-11-15 (Estimated)

PRIMARY OUTCOMES:
Phase 1b Adverse Events (AEs) | 2 years
  The incidence and severity of adverse events (AEs)
Phase 1b Dose-limiting toxicities | 28 days
  The DLT evaluation period is defined as the first 28 days of Cycle 1
Phase 2 Overall response rate (ORR) | 2 years
  Overall response rate (ORR) as defined by the International Myeloma Working Group (IMWG)

SECONDARY OUTCOMES:
Phase 1b Pharmacokinetic - AUC | 2 years
  Area under the curve of the GC012F (AZD0120) level
Phase 1b Pharmacokinetic - Cmax | 2 years
  Maximum GC012F (AZD0120) level
Phase 1b Pharmacokinetic - half-life | 2 years
  The elimination half-life of GC012F (AZD0120) level
Phase 1b Pharmacokinetic - Tmax | 2 years
  Time to reach Maximum GC012F (AZD0120) level
Phase 2: Adverse Events (AEs) | 2 years
  Further characterization of the safety of GC012F (AZD0120) by measuring the incidence and severity of AEs
Phase 1b and 2: Overall Response Rate (ORR) | 2 years
  ORR (sCR/CR/VGPR) is defined as the proportion of subjects who achieve sCR/CR/VGPR rate according to the IMWG criteria.
Phase 1b and 2: MRD negative rate | 2 years
  MRD negative rate as defined by the IMWG response criteria
Phase 1b and 2: Duration of response (DOR) | 2 years
  Duration of response (DOR) will be calculated among responders from the date of initial documentation of a response to the date of first documented evidence of progressive disease, as defined in the IMWG criteria, or death due to any cause, whichever occurs first.
Phase 1b and 2: PFS | 2 years
  Progression-free survival (PFS) defined as the time from the date of the initial infusion of GC012F to the date of first documented disease progression, as defined in the IMWG criteria, or death due to any cause, whichever occurs first.
Phase 1b and 2: OS | 2 years
  Overall survival (OS) is measured from the date of the initial infusion of GC012F to the date of the subject's death.

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - Research Site, Birmingham, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Aurora, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Iowa City, Iowa
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Rochester, Minnesota
  - Research Site, Omaha, Nebraska
  - Research Site, Hackensack, New Jersey
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, Stony Brook, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Charlottesville, Virginia
  - Research Site, Edmonds, Washington
  - Research Site, Seattle, Washington
  - Research Site, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: http://vivli.org